CLINICAL TRIAL: NCT01035060
Title: Role of Skeletal Muscle Blood in Muscle Regeneration and Sarcopenia
Brief Title: Blood Flow, Muscle Regeneration and Sarcopenia
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 37268
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2012-10

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum/Plasma; Skeletal Muscle; Adipose Tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Older Adult: Healthy Men and Women Over 70 Years of Age
- Young Adult: Healthy Men and Women Aged 18-30 Years

SUMMARY:
Due to the rapid aging of the population, sarcopenia is among the greatest challenges facing the health care system over the next quarter century. This age-related loss of skeletal muscle mass and strength directly contributes to the incidence of functional disability, thereby reducing independence and quality of life for the elderly. Despite increasing efforts to combat sarcopenia, its etiology remains incompletely described. Subsequently, limited progress has been made in developing comprehensive preventative and therapeutic strategies to combat the problem. A decreased ability to regenerate skeletal muscle fibers through the donation of skeletal muscle stem cells (satellite cells) is thought to contribute to sarcopenia. However, the upstream physiological mediators that regulate this impairment are poorly delineated.

Reduced muscle blood flow in advanced age appears to be a significant factor in reducing skeletal muscle regenerative capacity, but few data exist to confirm this hypothesis. Thus to test this hypothesis we aim to conduct a translational pilot trial which examines regeneration in both young and old adults. Furthermore, we aim to determine if muscle blood flow and satellite cell number are associated with muscle function. The central hypothesis of this proposal is that age-related declines in skeletal muscle angiogenesis and perfusion are significant causal factors in age-related losses of skeletal muscle mass. The specific aims and hypotheses of the project are as follows:

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-30 years
* Men and women aged > 70 years
* Body mass index < 35
* Willing and able to participate in all aspects of the study
* Sedentary to moderately active lifestyle <120 min physical activity/week < 30 min moderate aerobic exercise/week < 30 min resistance training/week OR Participates in regular structured exercise > 120 min/week
* Non-smoking

Exclusion Criteria:

* Active treatment for cancer, stroke (< 6 mo), peripheral vascular disease, coronary artery disease (myocardial infarction <6 mo), state III, IV Congestive Heart Failure, valvular heart disease, major psychiatric disease, severe anemia, liver or renal disease, diabetes, severe osteoarthritis, blindness or deafness, fracture in upper or lower extremity within the last 6 months, upper or lower extremity amputation, anticoagulant therapy (aspirin use is permitted), parkinsons disease
* Failure to give consent
* Anabolic medications (growth hormone or testosterone)
* High amounts of physical activity (i.e. running, bicycling etc > 120 min/week).
* Dementing illness
* Smoking
* Pregnant
* Significant cognitive impairment; Mini-Mental State (MMSE) exam < 24
* Statin Usage
* Excessive alcohol use (>2 drinks per day)
* Resting heart rate > 120 bpm
* Systolic blood pressure > 180 mmHg
* Diastolic blood pressure > 110 mmHg
* History of significant head injury
* Anticholinesterase inhibitor (such as Aricept)
* Contraindications to MRI (e.g. cardiac pacemaker, implanted cardiac defibrillator, aneurysm clip, claustrophobia, etc.)
* Current Use of Antidepressant Medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W. Buford, PhD, Principal Investigator — University of Florida
Locations (1):
- Aging and Rehabilitation Research Center, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2010 through December 2011, community-dwelling persons were recruited to participate through a variety of methods including media articles, direct mailings, newspaper announcements, and presentations to community groups.
Groups:
- Older Adults: Persons aged ≥ 70 years
- Young Adults: Persons aged 18-30 years
Period: Overall Study
Arm/Group | Older Adults | Young Adults
Started | 39 | 29
Completed | 15 | 15
Not Completed | 24 | 14
Not completed — Lost to Follow-up | 0 | 7
Not completed — Did not quality after 2nd screening | 14 | 1
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Older Adults | Young Adults | Total
Number analyzed (Participants) | 39 | 29 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 29 | 29
  >=65 years | 39 | 0 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 24 | 18 | 42
Region of Enrollment [Number; unit: participants]
  United States | 39 | 29 | 68

OUTCOME MEASURES:

1. Primary Outcome: Muscle Satellite Cells
Description: Change in the number of myonuclear cells identified as Pax7+ following contraction-induced skeletal muscle injury. Cells identified as Pax7+ by immunohistochemistry of skeletal muscle biopsy samples. Data adjusted for gender, physical activity level, and baseline satellite cell number.
Time Frame: Baseline, 2 days post-injury, 7 days post-injury
Measure: Mean (Standard Error); unit: Number of Pax7+ cells/muscle fiber
Groups:
- Older Adults: Age > 70 years
- Young Adults: Age 18-35 years
Arm/Group | Older Adults | Young Adults
Number analyzed (Participants) | 15 | 15
Number of Pax7+ cells/muscle fiber
  Adjusted Baseline | 3.2 (0.0) | 3.2 (0.0)
  Adjusted 2 days post-injury | 4.0 (.4) | 3.8 (0.4)
  Adjusted 7 days post-injury | 4.0 (0.3) | 3.7 (0.3)

ADVERSE EVENTS:
Time Frame: 14 months
Description: Data collected during study visits from September 2010 to December 2011
Arm/Group | Younger Adults | Older Adults
Serious Adverse Events (participants affected / at risk) | 0/29 | 2/39
Other Adverse Events (participants affected / at risk) | 6/29 | 7/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger Adults (N=29) | Older Adults (N=39)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) — Not as a result of the study
Hospitalization (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Participant was hospitalized for blood clots in both legs
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger Adults (N=29) | Older Adults (N=39)
Skeletal Muscle Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) — In response to exercise bout
Pain/Bruising (General disorders) | 4 (5) | 1 (1) — Following muscle biopsy
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Unrelated to study procedures
Broken Toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated to study procedures
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mild swelling (General disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Unrelated to study procedures
Minor Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No